CLINICAL TRIAL: NCT06717841
Title: Evaluation of Time-in-range and Glycemic Variability in Patients With Type 1 Diabates Mellitus and Celiac Disease With a Glycemic Monitoring Sensor
Brief Title: Metabolic Control and Glycemic Variability in Type 1 Diabetes and Celiac Disease
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CELTEC2020
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes Mellitis; Celiac Disease
Keywords: Type 1 Diabetes Mellitus; Celiac disease
MeSH Terms: conditions — Celiac Disease; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, retrospective study focused on differences of time-in-range and glycemic variability between a cohort of patients with both type 1 diabetes and celiac disease, and a cohort of patients with only type 1 diabetes.

DETAILED DESCRIPTION:
The study design provides for 2 cohorts of pediatric and adolescent patients using the continuous glycemic monitoring sensor. Cohort A consists of patients with type 1 diabetes and celiace disease, while cohort B consists of patients with only type 1 diabetes.

The primary aim of the study is to assess whether cohort A patients can achieve the same metabolic control and glycemic variability goals (expressed as Time-In-Range and glycemic Variability Coefficient) as cohort B patients.

The secondary aims are: assessing differences in Time-In-Range and glycemic Variability Coefficient between cohort A patients treated with multidaily injections, and those treated with continuous subcutaneous insulin infusion; assessing differences on total daily insulinic intake between cohort A and cohort B.

ELIGIBILITY:
Inclusion Criteria:

* patients < 18 years of age at enrollment;
* patients with type 1 diabetes onset since at least 1 year and celiac disease (COHORT A);
* patients only with type 1 diabetes onset since at least 1 year (COHORT B);
* using the continuous glycemic monitoring sensor;
* being on treatment with continuous subcutaneous insulin infusion or multidaily injections;
* obtaining informed consent from parents/legal guardian of pediatric patients.

Exclusion Criteria:

* patients with diabetes other than type1 diabetes;
* patients not using the glycemic monitoring sensor.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged < 18 years at enrollement with type 1 diabetes and celiac disease or with only type 1 diabetes, treated with continuous subcutaneous insulin infusion or multidaily injections and using the continuous glycemic monitoring sensor.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences on metabolic control between cohort A and B | in the 14 days prior to the most recent outpatient visit between February 2019 and February 2020
  time-in-range
Differences on glycemic variability between cohort A and B | in the 14 days prior to the most recent outpatient visit between February 2019 and February 2020
  glycemic variability coefficient

SECONDARY OUTCOMES:
Differences on metabolic control between patients on different therapeutic regimen | in the 14 days prior to the most recent outpatient visit between February 2019 and February 2020
  time-in-range
Differences on glycemic variability between patients on different therapeutic regimen | in the 14 days prior to the most recent outpatient visit between February 2019 and February 2020
  glycemic variability coefficient
Differences on total daily insulinic intake between cohort A and B | in the 14 days prior to the most recent outpatient visit between February 2019 and February 2020
  U/kg/die

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Maltoni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy